CLINICAL TRIAL: NCT03525041
Title: The Randomly Controlled Trial of Optimal Surgical Method for CAD Patients Combined Moderate Functional Ischemic Mitral Regurgitation
Brief Title: Mitral Valve Repair Combined Coronary Artery Bypass Grafting(CABG) Verus CABG Alone on Functional Ischemic Mitral Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Dong Ran, chief of ward No.11,cardiac surgery, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015217146; Z151100003915084 (Other Grant/Funding Number: Beijing Municipal Science and Technology Commission)
Record Dates: First submitted 2018-04-29; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Mitral Valve Insufficiency
MeSH Terms: conditions — Coronary Artery Disease; Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABG+mitral valve annuloplasty (Active Comparator): Participants will undergo CABG and mitral valve annuloplasty.
  Interventions: Procedure: CABG; Procedure: mitral valve annuloplasty
- CABG (Active Comparator): Participants will undergo CABG only.
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — CABG will be performed using standard surgical techniques. All procedures will be performed with cardiopulmonary bypass(CPB). Saphenous vein(SV)will be used as conduit but harvesting methods will not be prescribed, and utilization of the left internal mammary artery (LIMA) is recommended when a left anterior descending (LAD) graft is indicated. The technical details of bypass grafting will not be prescribed. Complete revascularization will be performed, judging by the surgical investigator.
Procedure: mitral valve annuloplasty — Surgical techniques for mitral valve annuloplasty may need to be adjusted at the discretion of the surgeon, as based on intra-operative findings that may not be previously recognized in the pre-operative evaluation.
  Arms: CABG+mitral valve annuloplasty

SUMMARY:
Coronary artery bypass grafting(CABG) is an effective procedure in treating severe coronary artery disease(CAD). Optimal surgical method for CAD patients with functional ischemic mitral regurgitation(FIMR) is still controversial. This study will evaluate the different effectiveness of CABG plus mitral valve annuloplasty versus CABG alone on patients with moderate FIMR.

DETAILED DESCRIPTION:
CAD is a severe health problem worldwide. It is a result of plaque buildup, and eventually leads to the reduction of blood supply on myocardium. CABG is one of the procedure to improve symptoms caused by myocardial ischemia. And it is especially effective in treating severe coronary artery disease.

FIMR is one of the most common complications of CAD. After acute myocardial infarction, FIMR will occur in 17%-55% patients, and 3%-19% of them will develop into moderate or severe MR eventually. FIMR is an important prognostic factor of CAD, the in-hospital mortality rate of patients with IMR is significantly higher in several studies. In patients with mild MR, CABG alone is enough to improve myocardial ischemia; however, in people with moderate mitral regurgitation, there is still a dispute on whether mitral valve annuloplasty is beneficial at the time of CABG. The purpose of this study is to determine the optimal surgical procedure of CAD patients combined moderate FIMR.

This study will compare the effectiveness of different surgical procedure on people with moderate FIMR by enrolling people with enrolling people with CAD who require CABG procedure and have moderate mitral regurgitation. At baseline study, a questionnaire will be assigned to undergo either CABG surgery of CABG plus mitral calve annuloplasty. Blood, urine and tissue samples will be collected after the surgery. All participants will be followed up at month 1,3,6,12, participants will take part in a medication history review, a physical examination, a blood collection to evaluate the brain natriuretic peptide and an echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

1. CAD that is amenable to CABG and a clinical indication for revascularization
2. Moderate mitral regurgitation in the judgment of the clinical site echocardiographer, quantitative guidelines as proposed would be: jet area between 4 cmsq to 8 cmsq, jet area/left atrial area ratio between 20% to 39%
3. Age ≥ 18 years
4. Mitral valve annuloplasty is applicable

Exclusion Criteria:

1. Organic mitral insufficiency caused by rupture of papillary muscle, rheumatic fever, degeneration or infectious endocarditis
2. Jet area of mitral valve cannot be evaluated by echocardiogram
3. In combination of other procedures such as surgery on tricuspid valve, aortic valve, congenital heart diseases or diseases of the thoracic arteries
4. Prior surgical or percutaneous mitral valve repair
5. Contraindication to cardiopulmonary bypass (CPB)
6. Clinical signs of cardiogenic shock at the time of randomization
7. Treatment with medication prior to the surgery
8. Severe, irreversible pulmonary hypertension in the judgment of the investigator
9. Evidence of cirrhosis or liver synthetic failure
10. Recent history of psychiatric disease (including drug or alcohol abuse) that is likely to impair compliance with the study, in the judgment of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular End Systolic Volume Index (LVESVI) | Measured at month 12

SECONDARY OUTCOMES:
Operative death | Measured during operation
In-hospital death | 1 year
  death during the time of hospitalization
Short-term complications | Measured within 1 week after operation
  Postoperative perivalvular leakage or heart failure
Rehospitalization | 1 year
  Re-hospitalization caused by heart failure or aggravated mitral regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Ran Dong, MD, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No